CLINICAL TRIAL: NCT07306130
Title: Consensus on Skin Care in Breast Cancer Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Venus Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: Breast Cancer-Venus
Record Dates: First submitted 2025-12-06; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Rejuvenation; Skin Care Dermocosmetics; Breast Cancer
Keywords: Dermocosmetics; skin care; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncodermatology-Focused Skincare: A cohort of dermatology and aesthetic medicine experts from the MENA region participating in a Modified Delphi process to develop consensus recommendations on Skin care in Breast Cancer.

SUMMARY:
Skin toxicity is one of the most common and impactful adverse effects of breast cancer treatment, affecting patients undergoing chemotherapy, targeted therapies, endocrine therapy, and radiotherapy. Current research and expert consensus highlight the importance of early, preventive, and gentle skin-care regimens to preserve barrier function and reduce treatment interruptions. Evidence supports the use of mild, fragrance-free cleansers, twice-daily emollient moisturization, and consistent broad-spectrum photoprotection throughout therapy. For radiation dermatitis, studies show that prophylactic moisturizers, silicone- or hydrofilm-based dressings, and short-course topical corticosteroids significantly reduce severity. Targeted therapies, particularly EGFR/HER2 inhibitors, require anticipatory management with barrier repair, topical anti-inflammatory agents, and oral antibiotics when papulopustular eruptions develop. Dermocosmetic products designed for sensitive or oncology-treated skin have demonstrated improvements in symptom burden and quality of life. Overall, the consensus emphasizes patient education, avoidance of irritants, multidisciplinary dermatologic-oncologic collaboration, and proactive rather than reactive care to effectively mitigate skin-related adverse events in breast cancer patients.

DETAILED DESCRIPTION:
Study Overview

This study is a non-interventional, observational expert consensus project designed to develop region-appropriate guidelines for skin care management in breast cancer patients undergoing systemic therapies, radiotherapy, or surgical treatment. Although numerous international guidelines address cancer-related skin toxicities, most are derived from Western populations and do not fully reflect regional differences in skin phototypes (Fitzpatrick III-VI), environmental factors, product availability, and care pathways common in the Middle East and North Africa (MENA) region. Because breast cancer patients frequently experience treatment-related dermatologic adverse events that affect quality of life and treatment adherence, a structured expert consensus is required to standardize preventive and therapeutic skin-care practices across oncology and dermatology settings.

Study Design

This study follows a Modified Delphi methodology, The Delphi process will include 2-3 iterative rounds:

Round 1 - Qualitative Item Generation

Experts will complete an open-ended questionnaire covering:

baseline skin-care recommendations (cleansing, moisturization, photoprotection); management of radiotherapy-induced dermatitis; chemotherapy- and targeted-therapy-related skin toxicities (xerosis, papulopustular rash, nail changes, photosensitivity); surgical wound and scar care; use of dermocosmetics and supportive products during cancer therapy; safety considerations for Fitzpatrick III-VI skin; contraindicated products or procedures (exfoliants, retinoids, lasers, waxing);

patient-education strategies; follow-up schedules and referral pathways; regional barriers (product availability, cultural factors, climate impact). Responses will undergo thematic analysis to produce structured statements.

Round 2 - Quantitative Consensus Rating

Panelists will rate the consolidated statements using a 9-point Likert scale (1 = inappropriate, 9 = appropriate), assessing clinical utility, safety, feasibility, and applicability to breast cancer care in the MENA region.

Optional Round 3

Only statements without clear consensus will undergo a third round. Experts will review anonymized group statistics (median, distribution spread) and re-rate remaining borderline items, allowing refinement of near-agreement topics.

Expert Panel Selection

Experts will be eligible if they meet at least two of the following criteria:

* ≥5 years of clinical experience in dermatology, oncology, or supportive cancer care;
* Recognized national or regional lecturer, trainer, or key opinion leader;
* Peer-reviewed publications in dermatology, oncology, supportive care, or cancer survivorship;
* Active practice within Egypt or other MENA countries.

The targeted panel size is 15-25 experts, ensuring representation across dermatology, radiation oncology, medical oncology, nursing, and survivorship care.

Statistical Analysis For each item, the following will be calculated: median, interquartile range, interpercentile range (IPR), IPR adjusted for symmetry (IPRAS), and the Disagreement Index. Items will be categorized by agreement level and summarized for publication. Subgroup analyses (e.g., GCC vs North Africa) may be performed.

Ethical Considerations This study does not involve patients, clinical interventions, or personal health information. Participation is voluntary. Expert responses are anonymized. No foreseeable risks are associated with participation, and the study qualifies as minimal-risk, non-interventional research.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Expertise: Must be a practicing healthcare professional (HCP) with a minimum of [e.g., 5-10] years of clinical experience in breast cancer management, supportive care, or oncology-related dermatology.
* Geographic and Practice Diversity: Representation from different geographical regions and practice settings (e.g., academic centers, community hospitals) to ensure broad applicability of the recommendations.

Availability and Willingness to Participate: Must formally agree to commit to the entire multi-round Delphi process (typically 2-4 rounds) within the specified timeline.

Exclusion Criteria:

* Inability or unwillingness to complete Delphi rounds.
* Lack of clinical experience with breast cancer patients.
* Industry representatives without direct clinical practice.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A purposively selected group of dermatology and aesthetic medicine experts from Egypt and the broader MENA region. Participants are clinicians with significant experience in skin care in breast cancer patients and are invited to contribute to a structured Modified Delphi process to develop regional consensus recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Achievement of Consensus on Skin Care in Breast Cancer patients | 6-12 weeks
  The final set of evidence-based and/or expert-supported statements, interventions, or practice recommendations for skin care in breast cancer patients that reach a pre-defined threshold of agreement among the expert panel.

CONTACTS AND LOCATIONS:
Locations (1):
- Venus Research Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Delphi studies do not collect patient data, medical records, biological samples, or identifiable clinical information. Experts only give opinions, not "IPD." Their responses are anonymized, and sharing identifiable expert-level responses is not required and often discouraged